CLINICAL TRIAL: NCT03936816
Title: The Implementation of Real-time PCR for Detection of Intrapartum GBS (Group B Streptococcus) Colonization as a Way to Reduce Antibiotic Prophylaxis Usage
Brief Title: The Implementation of Real-time PCR - Intrapartum GBS (Group B Streptococcus) Colonization to Reduce Antibiotic Prophylaxis
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Collaborators: Cepheid (Industry)
Responsible Party: Sponsor
Other Study IDs: CMC-19-0027-CTIL
Record Dates: First submitted 2019-04-08; First posted 2019-05-03 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: GBS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GBS screened positive: 150 patients that were screened positive by culture at 35-37 weeks gestational age.
  Interventions: Other: GBS vaginal double swab
- GBS unknown with risk factors: 150 patients that were not screened for GBS and have risk factors for GBS prophylaxis.
  Interventions: Other: GBS vaginal double swab

INTERVENTIONS:
Other: GBS vaginal double swab — The vaginal double swab will be assessed by two different lab tests: The first one for GBS culture on selective media after enrichment of 16h and the second swab by the Cepheid Xpert GBS Assay performed on the GeneXpert Dx system which is a qualitative in vitro diagnostic test designed to detect GBS DNA from vaginal swab specimens, using fully automated real-time polymerase chain reaction (PCR).

SUMMARY:
The implementation of real-time PCR for detection of intrapartum GBS (group B Streptococcus) colonization as a way to reduce antibiotic prophylaxis usage.

DETAILED DESCRIPTION:
The investigators intend to perform a cohort prospective trial in the delivery ward of CARMEL medical center. Pregnant women that are admitted to our ward and need to receive GBS (group B Streptococcus) prophylaxis either due to a positive GBS culture screen done at 35-37 weeks or by having risk factors for prophylactic antibiotic treatment (prolonged rupture of membranes, preterm delivery, GBS bacteriuria during current pregnancy) will be tested by a double vaginal swab (PCR and culture). Pregnant women that were screened positive at 35-37 weeks, those who had GBS bacteriuria during pregnancy and those who labor prematurely will be tested upon admission. Patients that have prolonged rupture of membranes (18 hours) will be tested by a double vaginal swab after 17 hours and prior to antibiotics administration.

All patient will be treated with GBS prophylactic antibiotics according to the culture screen done at 35-37 weeks or by risk factors (current protocol guidelines). Culture and PCR will be sent to the lab and the results will be revealed after delivery (the staff and patients will be blinded to the results of the culture and PCR until after delivery) in order to assess the number of patients that were treated with antibiotics unnecessarily.

The investigators intend to recruit 300 patients of which half will need antibiotics because of a positive culture at 35-37 weeks and half because of having risk factors. We decided to omit patients that will have fever during labor (a risk factor that necessitates GBS prophylaxis) because these patients will receive broad spectrum antibiotics anyway.

The vaginal double swab will be assessed by two different lab tests: The first one for GBS culture on selective media after enrichment of 16h and the second swab by the Cepheid Xpert GBS Assay performed on the GeneXpert Dx system which is a qualitative in vitro diagnostic test designed to detect GBS DNA from vaginal swab specimens, using fully automated real-time polymerase chain reaction (PCR).

ELIGIBILITY:
inclusion criteria:

* Pregnant patients that were screened positive by a culture at 35-37 weeks (those patients will be screened with a vaginal double swab upon admission to labor ward).
* Pregnant patients with GBS bacteriuria in current pregnancy (those patients will be screened with a vaginal double swab upon admission to labor ward).
* Pregnant patients in preterm labor before 37 weeks (those patients will be screened with a vaginal double swab upon admission to labor ward).
* Pregnant patients with prolonged rupture of membranes (those patients will be screened with a vaginal double swab after 17 hours and prior to antibiotics treatment).
* All patients have signed an informed consent.

Exclusion Criteria:

* Pregnant patients that do not want to participate in the study.
* Pregnant patients that fever is the risk factor for GBS prophylaxis.
* Pregnant patients that were screened negative by a culture at 35-37 weeks.
* Pregnant patient with PPROM (before 34 weeks).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: A cohort of 300 patient admitted to the labor ward in CARMEL medical center that need prophylactic antibiotics for GBS because of culture screen at 35-37 weeks or because of having risk factors.
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
intrapartum GBS PCR in patients that require GBS prophylaxis | The patients will be assessed once upon admission to labor room by having a double vaginal swab for GBS PCR and GBS culture
  The investigators intend to compare the number of patients that require GBS prophylaxis because they were screened positive (at 35-37 weeks) or have risk factors during labor (300 patients) to the number of patients that will be found positive on real time PCR upon admission to labor room. In that way the reduction (in percentage) for the need of GBS prophylaxis will be assessed.

SECONDARY OUTCOMES:
validity of GBS PCR | The patients will be assessed once upon admission to labor room by having a double vaginal swab for GBS PCR and GBS culture
  Each patient that will be recruited will be sampled vaginally by a double swab for PCR and culture for GBS. The investigators intend to compare the number positive results of PCR GBS to the number of positive culture results (which is considered gold standard) and in that way to determine the sensitivity and specificity of PCR for GBS.

CONTACTS AND LOCATIONS:
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No